CLINICAL TRIAL: NCT05833204
Title: Barbed Versus Standard Suture for Vaginal Cuff Closure After Total Laparoscopic Hysterectomy: a Randomized Controlled Trial
Brief Title: BARBED vs. STANDARD Suture for Colporrhaphy at the End of Laparoscopic Hysterectomy
Acronym: BARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Associate Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BARD
Record Dates: First submitted 2023-04-01; First posted 2023-04-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Vaginal Cuff Complications
Keywords: Laparoscopy; Hysterectomy; Vaginal cuff closure; Barbed sutures; Vaginal cuff complications; Vaginal cuff dehiscence

STUDY DESIGN:
Intervention Model Description: Multicenter, parallel arms, open-label, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeon will not be blinded. Conversely, patients and co-investigators who will assess study outcomes and perform patients' follow-ups will be masked regarding the allocation arm until the study's conclusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colporrhaphy with barbed absorbable suture (Experimental): The colporrhaphy will be performed using a 0-caliber barbed absorbable suture (V-Loc ™, Covidien, Medtronic)
  Interventions: Procedure: Laparoscopic colporrhaphy with 0-caliber barbed absorbable suture
- Colporrhaphy with standard absorbable suture (Active Comparator): The colporrhaphy will be performed using a standard 0-caliber absorbable suture made of a coated braided thread (Vicryl; Ethicon Inc, Sommerville, NJ)
  Interventions: Procedure: Laparoscopic colporrhaphy with standard 0-caliber absorbable suture

INTERVENTIONS:
Procedure: Laparoscopic colporrhaphy with 0-caliber barbed absorbable suture — After the total laparoscopic hysterectomy, the colporrhaphy will be performed using a 0-caliber barbed absorbable suture (V-Loc ™, Covidien, Medtronic)
  Arms: Colporrhaphy with barbed absorbable suture
Procedure: Laparoscopic colporrhaphy with standard 0-caliber absorbable suture — After the total laparoscopic hysterectomy, the colporrhaphy will be performed using a 0-caliber absorbable suture made of a coated braided thread (Vicryl; Ethicon Inc, Sommerville, NJ)
  Arms: Colporrhaphy with standard absorbable suture

SUMMARY:
Hysterectomy is one of the most common surgical procedures performed worldwide, with more than 400,000 hysterectomies performed annually in the United States. As a consequence, even uncommon complications can affect large numbers of patients. Among potentially life-threatening events, vaginal cuff dehiscence complicates 0.14-1.38% of procedures, and any vaginal cuff complications (dehiscence, hematoma, bleeding, infection) are estimated to affect 4.7-9.8% of patients. In this scenario, any preventive strategy can provide clinically relevant benefits. Regarding colporrhaphy, only the adoption of a laparoscopic approach instead of a vaginal approach is supported by high-quality evidence. Our group demonstrated that the laparoscopic closure of the vaginal cuff after total laparoscopic hysterectomy reduces the incidence of vaginal cuff complications.

Among other potentially effective interventions, the use of barbed sutures was associated with a lower incidence of vaginal cuff dehiscence than the standard suture. In a recent meta-analysis, the use of barbed sutures has been associated with a pooled incidence of vaginal cuff dehiscence of 0.4% versus 2% after a traditional vaginal suture. However, this evidence is limited because most pooled studies were retrospective, and only two were randomized controlled trials. Moreover, these two randomized controlled trials had a very small sample size and were not powered to detect clinically relevant differences. On that basis, despite the promising utility of barbed sutures for vaginal cuff closure after total laparoscopic hysterectomy, the choice of the type of suture is not evidence-based but still guided by personal opinions, as well as by the preference and habits of the operators.

Therefore, this study aims to investigate whether the laparoscopic vaginal cuff closure with barbed suture determines a lower incidence of vaginal cuff dehiscence and complications than conventional sutures after total laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total laparoscopic hysterectomy
* Surgery performed for the treatment of benign pathology
* Age > 18 years
* Surgery performed by laparoscopy
* Signature of informed consent

Exclusion Criteria:

* Patients undergoing emergent surgery
* Patients candidates for hysterectomy for oncological indication
* Patients who underwent previous radiation therapy
* Patients allergic to the suture material used in the study
* Patients unable to express adequate informed consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1614 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal cuff dehiscence | 30 days after surgery
  Any partial or total separation of the vaginal cuff
Vaginal cuff dehiscence | 90 days after surgery
  Any partial or total separation of the vaginal cuff

SECONDARY OUTCOMES:
Vaginal cuff complications | 30 days after surgery
  Hematoma, abscess, infections, bleeding, resuture of the vaginal cuff
Vaginal cuff complications | 90 days after surgery
  Hematoma, abscess, infections, bleeding, resuture of the vaginal cuff
Hospital stay | From the date of hospital admission to the date of hospital discharge.
  Days of hospitalization from the day of admission to the day of discharge.
Operative time | During surgery
  Time between first incision and skin closure
Intraoperative blood loss | During surgery
  Total blood aspirate during the surgical procedure
30-day post-surgical morbidity | 30 days after surgery
  Perioperative (intraoperative and postoperative) complications graded based on the Clavien-Dindo classification
Quality of life index | 90 days after surgery
  The Short Form 12 Health Survey (SF-12) investigates 8 different health aspects. Physical activity, role and physical health, role and emotional state, and mental health are measured by two questions. The SF-12 scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Sexual function | 90 days after surgery
  The female sexual function index (FSFI) consists of 19 multiple-choice items that assess female sexual functioning based on 6 domains: desire, arousal, orgasm, pain, sexual satisfaction, and lubrication. The total score ranges from 0 to 36, with 26.55 as the cut-off suggesting the presence of sexual dysfunction. The higher the score, the better the sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Principal Investigator — Universita di Verona; Simone Garzon, MD, Principal Investigator — Universita di Verona; Pier Carlo Zorzato, MD, Principal Investigator — Universita di Verona
Locations (1):
- AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uccella S, Zorzato PC, Kho RM. Incidence and Prevention of Vaginal Cuff Dehiscence after Laparoscopic and Robotic Hysterectomy: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2021 Mar;28(3):710-720. doi: 10.1016/j.jmig.2020.12.016. Epub 2021 Jan 5. PMID 33348012
- [Background] Uccella S, Malzoni M, Cromi A, Seracchioli R, Ciravolo G, Fanfani F, Shakir F, Gueli Alletti S, Legge F, Berretta R, Corrado G, Casarella L, Donarini P, Zanello M, Perrone E, Gisone B, Vizza E, Scambia G, Ghezzi F. Laparoscopic vs transvaginal cuff closure after total laparoscopic hysterectomy: a randomized trial by the Italian Society of Gynecologic Endoscopy. Am J Obstet Gynecol. 2018 May;218(5):500.e1-500.e13. doi: 10.1016/j.ajog.2018.01.029. Epub 2018 Feb 2. PMID 29410107